CLINICAL TRIAL: NCT06306391
Title: Physiologically Based Pharmacokinetic Modelling of Intravenous and Intranasal Formulations of Naloxone in Healthy Volunteers.
Brief Title: Pharmacokinetics of Intravenous and Intranasal Formulations of Naloxone in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IMIMFCTL/NLX_1
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous naloxone (Experimental): Assignment of treatment is sequence randomized. One single intravenous dose on Period 1 Day 1 and one single intranasal dose administered in supine position on Period 2 Day 1 or vice versa.
  Intravenous naloxone as IV bolus using external infusion pump will be administered to subjects after at least 8 hours (10 hours +/- 2 hours) of fasting conditions.
  Interventions: Drug: Intravenous naloxone
- Intranasal naloxone (Experimental): Assignment of treatment is sequence randomized. One single intravenous dose on Period 1 Day 1 and one single intranasal dose administered in supine position on Period 2 Day 1 or vice versa.
  One intranasal dose of naloxone nasal spray will be administered in one nostril following the instructions described in the protocol after at least 8 hours (10 hours +/- 2 hours) of fasting conditions.
  Interventions: Drug: Intranasal naloxone

INTERVENTIONS:
Drug: Intravenous naloxone — Nyoxid 1.8 mg nasal spray, solution in single-dose container. Study drugs (naloxone nasal spray and naloxone intravenously) will be administered in 8 subjects in two sequences in fasting conditions (10 hours pre-dose and 4 hours post dose): Intranasal -> washout period ->intravenous (n=4) and Intravenous ->washout period -> intranasal (n=4).
  Other Names: Intravenous - washout - intranasal
  Arms: Intravenous naloxone
Drug: Intranasal naloxone — Naloxone Kern Pharma 1 mg in total (from 0.4 mg/mL injectable solution). Study drugs (naloxone nasal spray and naloxone intravenously) will be administered in 8 subjects in two sequences in fasting conditions (10 hours pre-dose and 4 hours post dose): Intranasal -> washout period ->intravenous (n=4) and Intravenous ->washout period -> intranasal (n=4).
  Other Names: Intranasal - washout - intravenous
  Arms: Intranasal naloxone

SUMMARY:
This is a phase I interventional clinical trial and the aim will be to characterize the PK and PD of two formulations of naloxone (intranasal and intravenous) in healthy subjects, which will be used to verify/validate nasal-CNS-PBPK (Physiologically Based Pharmacokinetic) model predictions following intranasal dosing.

DETAILED DESCRIPTION:
Naloxone is a semisynthetic morphine derivative and is a specific opioid antagonist that acts competitively at opioid receptors. It reveals very high affinity for the opioid receptor sites. Naloxone does not possess the "agonistic" or morphine-like properties characteristic of other opioid antagonists. In the absence of opioids or agonistic effects of other opioid antagonists, it exhibits essentially no pharmacologic activity. Naloxone has not been shown to produce tolerance or cause physical or mental dependence. Intranasally administered naloxone has been demonstrated to be rapidly absorbed, as evidenced by very early appearance (as early as 1 minute after administration) of the active substance in systemic circulation. A study investigating intranasal naloxone (Nyxoid™) at doses of 1, 2, 4 mg (MR903-1501) shows that the median (range) tmax associated with intranasal administration of naloxone was 15 (10, 60) minutes for 1 mg, 30 (8, 60) minutes for 2 mg and 15 (10, 60) minutes for 4 mg intranasal doses. Onset of action following intranasal administration can reasonably be expected to occur in each individual before the tmax is reached.

The half value duration (HVD) for intranasal administration were longer than for intramuscular administration (intranasal, 2 mg, 1.27h, intramuscular, 0.4 mg, 1.09h) from which we can infer a longer duration of action of naloxone given by the intranasal rather than the intramuscular route. The overall aim is to develop a physiologically based pharmacokinetic (PBPK) model for drug release, disposition and dissolution following intranasal drug delivery. Following delivery, drug release from the formulations and disposition in the nasal cavity will be described. The model will also account for drug transport through epithelial tissue and mucociliary clearance. Predicted local brain and systemic PK will therefore be linked to drug release, dissolution, and disposition in the brain and the rest of the body. In vitro permeability, transporter kinetic and proteomics data from the olfactory region, as well as published clinical data following intravenous and intranasal delivery will be used to support this. Integration of all these processes in a dynamic model will help to disentangle different kinetic process which contribute to this complex system, which will help us to explore the interplay between various processes. Intranasal: 1.8 mg nasal spray, solution in single-dose container. Intravenous: 1 mg in total (from 0.4 mg/mL injectable solution) Doses selected, in the low range of those tested previously in clinical opioid overdose situations, were already tested experimentally in a bioavailability study in healthy subjects comparing the two routes of administration of naloxone that will be evaluated in the protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female volunteers according to physical examination, vital signs (blood pressure, heart rate and body temperature), ECG and safety laboratory parameters and results should be within normal ranges or considered as non-clinically relevant by the investigator.
2. Age ≥ 18 and ≤ 55 years.
3. Body mass index (BMI) ≥ 18 and ≤ 30.
4. Able/willing to be compliant with the study restrictions.
5. Able to read Spanish and adhere to study requirements.
6. Signed informed consent prior to any study-mandated procedure.

Exclusion Criteria:

1. - Life-time substance use disorders (SUD) according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5).
2. - Consumption of prescribed opiates (in the last 6 months).
3. - Smoking.
4. - History of or ongoing clinically relevant diseases or conditions.
5. - Being under any administrative or legal supervision.
6. - Pregnancy and breastfeeding
7. - Positive blood or urine test for drugs of abuse or alcohol breath test prior to study drug administration.
8. - Life-time history of mental diseases.
9. - History of anxiety or depression not completely recovered within 12 months prior to study drug administration, as assessed by the Dual Diagnosis Screening Interview (DDSI).
10. - Any other clinically relevant disease or condition that in the judgment of the investigator might interfere with the subject's ability to comply with study procedures or requirements and/or bias the interpretation of the study results and/or jeopardize the subject's safety.
11. - Ongoing gastrointestinal diseases or history of gastrointestinal surgery affecting absorption.
12. - Subjects with a clinically significant disease within one month prior to study drug administration.
13. - Any clinically relevant findings in physical examination, vital signs, 12-lead ECG and safety laboratory parameters.
14. - Positive hepatitis or HIV test.
15. - Known hypersensitivity to any drug or drug excipients.
16. - Use of drugs known to induce or inhibit hepatic drug metabolism (e.g., cimetidine) within one month prior to study administration or during the study and use of citrus juice during the study.
17. - Any prescription or over-the-counter (OTC) product including herbal, homeopathic, vitamins, minerals and nutritional supplements within one week prior to study drug administration.
18. - Intake of foods or beverages containing xanthine (more than 5 units of coffee, tea or cola drinks per day).
19. - Donation of blood or plasma within one month prior to study drug administration or transfusion of blood or plasma for medical/surgical reasons or intention to donate blood or plasma within one month after study drug administration.
20. - History of inadequate venous access and/or experience of difficulty donating blood.

    * Subject included in a clinical study within 3 months prior to study drug administration.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Effects of naloxone on heart rate (HR). | Up to 24 hours.
Effects of naloxone on systolic and diastolic blood pressure (BP). | Up to 24 hours.

SECONDARY OUTCOMES:
Effects of naloxone on plasma cortisol at visit 1 and visit 4. | Up to 24 hours.

OTHER OUTCOMES:
Adverse effects. | Up to 24 hours.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital del Mar Research Institute, Barcelona
  - IMIM (Hospital del Mar Medical Research Institute), Barcelona